CLINICAL TRIAL: NCT05204433
Title: Correlation Between Methylation Site of SFRP1 Gene Promoter and Colorectal Cancer and Adenoma
Brief Title: Correlation Between SFRP1 and Colorectal Cancer and Adenoma
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Jie Liang, Professor, Xijing Hospital of Digestive Diseases
Other Study IDs: XJLJ-Fecal-adenoma
Record Dates: First submitted 2022-01-11; First posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Early Diagnosis of Colorectal Cancer and Adenoma
MeSH Terms: conditions — Adenoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- normal control: healthy volunteers
  Interventions: Other: no intervention
- adenoma: pathologically reported colorectal adenoma
  Interventions: Other: no intervention
- colorectcal cancer: pathologically reported colon cancers
  Interventions: Other: no intervention
- High risk group: pathologically reported inflammatory bowel diseases

INTERVENTIONS:
Other: no intervention — no intervention
  Groups: adenoma; colorectcal cancer; normal control

SUMMARY:
In summary, our study demonstrated the methylation sites of SFRP1 gene promoter in patients with colorectal cancer and adenoma and found SFRP1_16_17_18 CpG site was good performance as a diagnostic marker of colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* consecutive adult patients undergoing an outpatient endoscopy and histopathologically diagnosed as colorectal cancer or adenoma. Also, healthy individuals were invited to be enrolled.

Exclusion Criteria:

* Lynch syndrome
* Familial adenomatous polyposis
* MUTYH associated polyposis
* Peutz-Jeghers syndrome
* Juvenile polyposis syndrome
* Serrated polyposis syndrome

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: consecutive adult patients undergoing an outpatient endoscopy
Sampling Method: Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2019-01-05 (Actual); Primary Completion 2022-02-20 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
effectiveness of methylation markers from stool samples | 3 years
  assess the effectiveness of methylation markers from stool samples in colon cancer patients, colorectal adenoma patients, compared with normal volunteers

SECONDARY OUTCOMES:
assess the capacities of RF model in screening potential clinical biomarkers. | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Jie Liang, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided